CLINICAL TRIAL: NCT01760785
Title: A Double Blind Trial of Divalproex Sodium for Affective Lability and Alcohol Use Following Traumatic Brain Injury
Brief Title: Valproate for Mood Swings and Alcohol Use Following Head Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0582; PT075168 (Other: Department of Defense)
Record Dates: First submitted 2012-11-08; First posted 2013-01-04 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Traumatic Brain Injury (TBI); Alcoholism
Keywords: Veterans; Traumatic Brain Injury(TBI); Alcoholism
MeSH Terms: conditions — Brain Injuries, Traumatic; Alcoholism | interventions — Valproic Acid; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- divalproex sodium (Active Comparator)
  Interventions: Drug: divalproex sodium
- sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: divalproex sodium — Doses will be given in 250mg increments and titrated over the first four days of study until a starting dose of 750 mg is reached. The Study Oversight Team, who is not involved in any clinical visits, will be un-blinded to study drug assignment and will have plasma concentration results and adverse event reports available to them. If a subject has no adverse events and is not at therapeutic level as indicated by the blood levels, the Study Oversight Team may inform the research pharmacy to increase the dose by 1 tablet of 250 mg to 1000 mg per day. The Study Oversight Team may also inform the research pharmacy to reduce the daily dosage back down to 750 mg per day if plasma concentrations or adverse events become intolerable. The maximum dose for the purpose of this study will be 1250 mg daily and the minimum dose will be 750 mg daily. Subjects who cannot tolerate the minimum dose will be excluded from any further study participation.
  Arms: divalproex sodium
Drug: Placebo — Doses will be titrated over the first four days of study in the same manner as the active study drug. After titration, the research pharmacy may increase the dose by 1 tablet per day, in the same fashion that the active drug may be adjusted, so that the participant and clinical team remain blinded to the drug assignment. The research pharmacy may also reduce the daily dosage back down by one tablet per day for the same reason.
  Other Names: sugar pill
  Arms: sugar pill

SUMMARY:
Successful treatment of traumatic brain injury (TBI)-induced mood lability may reduce or eliminate drinking behaviors in persons with alcohol abuse/dependence (AA/D) and affective lability following TBI. Observed clinically, the symptoms of poorly regulated affective expression of AA/D+TBI patients who reach alcohol abstinence do not appear to be those of an idiopathic mood or anxiety disorder. These symptoms do not present the severity or the same natural courses as do Major Depressive Disorder, Bipolar Illness, or Anxiety Disorder, for example. Instead, both symptoms and course appear more characteristic of the sustained affect lability often observed following TBI. This observation suggests that TBI survivors represent a patient group for whom treatment of neuropsychiatric symptoms following TBI may alleviate both TBI-related affect lability and also heavy ethanol use by treating the condition that is contextually related to excessive alcohol use.

Based on this concept of consequently treating AA/D through the management of post-TBI affective lability, this study was conducted observing the efficacy of divalproex sodium on the severity of affective lability and AA/D in persons suffering from a moderate TBI. Divalproex sodium has been shown to ameliorate mood disorders, even in those with substance abuse problems. This drug has also shown positive results as an alternate medication to benzodiazapines in the treatment of alcohol withdrawal, significantly reducing the progression of withdrawal symptoms in patients.

DETAILED DESCRIPTION:
Despite the body's natural healing during the first year after a head injury, many veterans who have suffered even mild brain injuries find themselves easily upset or fearful as they go about their daily lives. While these reactions to the world around them were easily managed before the head injury, they now occur with little or no interruption and are exceedingly difficult to manage. Such reactions include a sense of always being upset or fearful that often makes it difficult to get along with family members, friends, coworkers, and employers. This may lead to broken marriages, unemployment, and even homelessness.

Some people with head injuries try to manage their unmanageable moods by drinking alcohol because it can create a sense of calm. However, alcohol's actions are short in duration. Most find that they have to drink more and more for a similar calming effect, and they soon become dependent on alcohol. This makes working and being part of their families even more difficult.

To treat the unmanageable mood, we tried a medicine called valproate, one that eases mood problems in people without head injury. We gave valproate to head injured persons with mood problems in a "non-blinded" study where both the doctor and the patient knew that the medicine was valproate and both were optimistic that it would work. In a small sample of eighteen people, 85% found mood relief and most of those either stopped drinking alcohol or drank much less than before. However, this might have been because both the doctor and patient were hopeful that the medication would make the patient feel better or because the medicine actually worked.

The only way to know for sure if the medicine works is to perform a study in which people receive either valproate or a sugar pill while neither they nor their doctor know which one they are taking. This is called a double blind study, as proposed here, and will involve nearly three times as many head injured persons as the first study.

If it is successful, the new study will show that valproate treatment helps head injured people manage their moods and allows them to return to families, friends, and work. It will also show that they drink alcohol less or not at all, improving their health even further. Then doctors will know that they can use this medicine for large numbers of people who suffer from head injury and help them to lead normal lives. If the outcome of the study shows that the medicine works well, doctors can then use this medicine to treat people with head injury immediately after the study results are published.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* history of closed-head traumatic brain injury (TBI) at least one year prior to enrollment
* symptoms of affective lability such as mood swings, irritability, frustration and anxiety
* currently using alcohol

Exclusion Criteria:

* history of Axis I bipolar disorder or anxiety disorder prior to the TBI
* skull opened either surgically or traumatically
* history of stroke
* current diagnosis or past history of major psychosis as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
* active liver disease
* evidence of the alcohol amnesic syndrome
* history of seizure disorder other than those caused by ethanol withdrawal
* any type of dementia
* current suicidal/homicidal ideations
* symptomatic thiamine, folate or Vitamin B-12 deficiency
* HIV positive
* any medical conditions that would constitute contraindications to treatment with divalproex sodium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2014-08 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Beresford, MD, Principal Investigator — Denver Veteran's Affairs Medical Center
Locations (1):
- Denver Veteran's Affairs Medical Center, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between in December 2008 and was completed in May 2014. Participants were recruited from the local VA medical center and the surrounding area. Recruitment included television advertisements, bus banners, flyers distribution, hospital signage, and word of mouth. 637 participants were initially screened via telephone.
Pre-assignment Details: Screening was done in two phases: telephone and in-person. Telephone screening included questions about the severity of the traumatic brain injury (TBI), substance use history, mood lability, medical and psychiatric history, and availability of proxy reporter. The in-person phase included screening for exclusionary cognitive or physical impairment.
Period: Overall Study
Arm/Group | Divalproex Sodium | Sugar Pill
Started | 23 | 27
Completed | 23 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Divalproex Sodium | Sugar Pill | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 27 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.99) | 45.3 (9.66) | 45.7 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Severity of Affective Lability Based on Shortened Agitated Behavior Scale
Description: Severity of affective lability was measured using a shortened version of the Agitated Behavior Scale (ABS). The ABS is used to assess the nature and extent of present agitation. Eight items from the 14-item scale were used, which measured the presence and severity of various affective lability symptoms including: short attention span, impulsivity, uncooperative behavior, violent tendencies, restlessness, rapid or excessive talking, sudden changes in mood, and easily initiated or excessive crying and/or laughter. Each of the eight items was scored using a 1-4 Likert scale, where 1 stands for absence of symptom and 4 stands for presence to an extreme degree. The minimum possible score for this measure was 8, and the maximum possible score was 32. Due to the nature of the measure, a lower score indicated less severe affective lability, while conversely higher scores indicated more severe affective lability. The mean of scores for weeks 2 through 8 for each group were reported.
Time Frame: Weeks 2 through 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Divalproex Sodium | Sugar Pill
Number analyzed (Participants) | 23 | 26
units on a scale | 9.22 (0.18) | 9.39 (0.25)

2. Secondary Outcome: Frequency of Alcohol Use
Description: Frequencies of alcohol use/misuse will be measured weekly utilizing the Timeline Followback assessment. Participants will also be given an alcohol breath test at every clinic visit.
Time Frame: Weeks 1-10
Measure: Mean (Standard Deviation); unit: standard drinks/day
Arm/Group | Divalproex Sodium | Sugar Pill
Number analyzed (Participants) | 23 | 26
standard drinks/day | 0 (0) | 0 (0)

ADVERSE EVENTS:
Arm/Group | Divalproex Sodium | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/27
Other Adverse Events (participants affected / at risk) | 0/23 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No